CLINICAL TRIAL: NCT01209988
Title: A Prospective Randomized Study Examining the Impact of Tamsulosin on Voiding Patterns Following Early Catheter Removal After Robot-Assisted Laparoscopic Radical Prostatectomy
Brief Title: Impact of Tamsulosin on Voiding Patterns Following Early Catheter Removal After Robot-assisted Laparoscopic Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Choung-Soo Kim/professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMC_UR_010
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Prostatic Neoplasms, Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamsulosin 0.4mg (Experimental): Perioperative tamsulosin 0.4mg daily
  Interventions: Drug: tamsulosin 0.4mg
- Control (Placebo Comparator): No medication
  Interventions: Other: No medication

INTERVENTIONS:
Drug: tamsulosin 0.4mg — perioperative tamsulosin 0.4mg daily for three weeks
  Arms: Tamsulosin 0.4mg
Other: No medication — No medication
  Arms: Control

SUMMARY:
To date, there is a lack of consensus concerning the optimal timing for removal of the urethral catheter, its related complications, the effectiveness in prophylactic drug use to reduce complication, and the patient reported outcomes (quality of life) after robot-assisted laparoscopic prostatectomy (RALP). The purpose of this study is to determine the impact of tamsulosin on voiding patterns following early urethral catheter removal after RALP for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have localized or locally advanced prostate cancer
* Patients must receive robot assisted laparoscopic radical prostatectomy
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Patients must not have a history of treatment with alpha blockers within 4 weeks
* Patients must not have previously undergone transurethral resection, laser therapy, or other surgery of the prostate
* Patients must not have previously been diagnosed with neurogenic bladder
* Patients must not have hypersensitivity to trial drug or other alpha-blockers
* Patients must not have the participation of other clinical trial within the past 3 months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of acute urinary retention | within the 30 days after surgery

SECONDARY OUTCOMES:
Patient reported outcomes | 20 days after surgery (plus or minus 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Choung-Soo Kim, M.D., Principal Investigator — Department of Urology, Asan Medical Center, Seoul, Korea
Locations (1):
- Asan Medical Center, Seoul, South Korea